CLINICAL TRIAL: NCT05981157
Title: Anrotinib Combined With Tirelizumab in First-line Treatment of Recurrent/Metastatic Nasopharyngeal Carcinoma
Brief Title: Anrotinib and Tirelizumab in First-line Treatment of RM-NPC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan People's Hospital, Guangdong, China (Other)
Responsible Party: Principal Investigator, Gui-Qiong Xu, Deputy director of Radiotherapy department for Nasopharyngeal and Head and Neck Tumors, Zhongshan People's Hospital, Guangdong, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZSCPH-001
Record Dates: First submitted 2023-05-16; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: nasopharyngeal carcinoma; Immunotherapy; Molecular Targeted Therapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anrotinib plus Tirelizumab arm (Experimental): Subjects receive anrotinib plus tirelizumab
  Interventions: Drug: Anrotinib plus Tirelizumab

INTERVENTIONS:
Drug: Anrotinib plus Tirelizumab — Subjects receive Anrotinib, 10mg, QD and Tirelizumab, 200mg, D1, Q3W. Treatment was continued until confirmed disease progression, death, unacceptable toxicity, withdrawal of consent, or investigator decision.

SUMMARY:
This is a prospective phase II clinical trial to evaluate the efficacy and safety of Anrotinib and Tirelizumab as a first-line treatment in patients with advanced recurrent or metastatic nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Had histopathologically confirmed nonkeratinizing recurrent/metastatic NPC (AJCC, 8th; the metastatic tissue biopsy is preferred, not necessary; locoregional recurrent lesion unfit for local treatment).
2. Subjects enrolled must have measurable lesion(s) according to response evaluation criteria in solid (RECIST) v1.1.
3. ECOG performance status of 0～2
4. Life expectancy more than 12 weeks.
5. unable or unwilling to undergo chemothraphy
6. Able to understand and sign an informed consent form (ICF).

Exclusion Criteria:

1. Uncontrolled clinically significant medical condition, including but not limited to the following: Hypertension that cannot be reduced to the normal range after antihypertensive drug congestive heart failure (New York Health Authority Class > 2), unstable angina, myocardial infarction within the past 12 months, clinically significant supraventricular arrhythmia or ventricular arrhythmia requiring treatment or intervention;
2. Known history of hypersensitivity to any components of the Tirelizumab formulation or other monoclonal antibodies ;
3. Diagnosed with other malignant tumors.
4. Subjects with any active autoimmune disease or history of autoimmune disease, or history of syndrome that requires systemic steroids or immunosuppressive medications, including but not limited to the following: rheumatoid arthritis, pneumonitis, colitis (inflammatory bowel disease), hepatitis, hypophysitis, nephritis, hyperthyroidism, and hypothyroidism, except for subjects with vitiligo or resolved childhood asthma/atopy. Subjects with the following conditions will not be excluded from this study: asthma that requires intermittent use of bronchodilators, hypothyroidism stable on hormone replacement, vitiligo, Graves' disease, or Hashimoto's disease. Additional exceptions may be made with medical monitor approval;
5. Subjects with medical condition affecting oral drug absorption, such as dysphagia, chronic diarrhea and intestinal obstruction.
6. Active bleeding, ulcer, intestinal perforation, major surgery in the previous month; Patients with tumors close to the internal carotid artery or other large vessels, thus at risk of massive bleeding.
7. The laboratory test values within 7 days before enrollment do not meet the relevant standards.
8. Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids. Doses 10 mg/day prednisone or equivalent are prohibited within 4 weeks before study drug administration. Note: corticosteroids used for the purpose of IV contrast allergy prophylaxis are allowed;
9. History of immunodeficiency including seropositivity for human immunodeficiency virus (HIV), or other acquired or congenital immune-deficient disease; active tuberculosis (TB), anti-TB treatment is ongoing or within 1 year prior to screening; Evidence of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection or risk of reactivation based on institutional guidelines and tests. Testing may include the following: HBV DNA, HCV RNA, hepatitis B surface antigen, or anti-Hepatitis B core antibody.
10. Subjects with comorbidities with long-term immunosuppressive drug therapy, or with systemic or local use of immunosuppressive doses of corticosteroids.
11. Subjects who underwent anti-PD-1 /PD-L antibody or anti-CTLA-4 antibody (or any other antibody acting on T cell synergistic stimulation or checkpoint pathway) and anti-angiogenic drugs.
12. Received any anti-infective vaccine (e.g. influenza vaccine, varicella vaccine, etc.) within 4 weeks prior to enrollment.
13. Any other medical (eg, pulmonary, metabolic, congenital, endocrinal, or CNS disease), psychiatric, or social condition deemed by the investigator to be likely to interfere with a subject's rights, safety, welfare, or ability to sign informed consent, cooperate, and participate in the study or would interfere with the interpretation of the results;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 1 year
  Defined as the proportion of patients whose tumors shrink to complete response (CR) or partial response (PR) and remain for a certain period of time according to RECIST 1.1

SECONDARY OUTCOMES:
The proportion of patients who achieved disease control | 1 year
  Defined as the proportion of subjects who achieve CR+PR+stable disease (SD) for at least 4 weeks according to RECIST 1.1.
The proportion of patients who achieved clinical benefit | 1 year
  Defined as maintaining the efficacy of CR+PR+SD for at least 6 months according to RECIST 1.1.
Duration of response | 1 year
  Defined as the time from the first assessment of CR and PR to the first assessment of PD or death caused by any cause according to RECIST 1.1.
progression-free survival | 1 year
  Defined as the period from the start of enrollment until disease progression or death from any cause.
Adverse events | 1 year
  NCI-CTC5.0 standard was adopted, and the safety was assessed mainly by clinical laboratory tests, ECOG-PS score, physical examination, electrocardiogram, and adverse event results.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan City People's Hospital, Zhongshan, Guangdong, China